CLINICAL TRIAL: NCT03573856
Title: Reducing Diabetes Risk Factors in American Indian Children: Tribal Turning Point
Acronym: TTP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17-1306; R01DK115434 (NIH)
Record Dates: First submitted 2018-05-21; First posted 2018-06-29 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Overweight/Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Health; Safety

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Living (Active Comparator): Three component behavioral intervention consisting of group-based classes, individual motivational interviewing-based sessions, and resource toolbox
  Interventions: Behavioral: Active Living
- Health and Safety (Placebo Comparator): One component health and safety program consisting of group classes
  Interventions: Other: Health and Safety

INTERVENTIONS:
Behavioral: Active Living — Participants will be provided with education and support for diet and lifestyle modification related to healthy eating and active living.
  Arms: Active Living
Other: Health and Safety — Participants will be provided with education related to general health and safety topics.
  Arms: Health and Safety

SUMMARY:
This study will evaluate a behavioral intervention designed to reduce risk factors for type 2 diabetes in American Indian youth aged 7-10 years.

DETAILED DESCRIPTION:
The objectives of tis study are to rigorously evaluate the effect of Tribal Turning Point (TTP) on diabetes risk factors in Native youth. The investigators will enroll up to 360 youth who are aged 7-10 years, overweight/obese (BMI >85th percentile), self-identify as American Indian, and have >1 parent/primary caregiver willing to actively participate in the program. Within each community, youth will be randomized to the TTP program or a general health and safety control program. The multi-component TTP intervention is a youth-centered adaptation of the Diabetes Prevention Program designed to reduce diabetes risk factors by improving activity and dietary behaviors. Informed by the pediatric weight management literature, the 12-month intervention includes 12 active learning group classes, 7 individual youth/parent motivational interviewing counseling sessions, and community-specific resource toolboxes. In this trial, the investigators will assess the effect of TTP on anthropometric, metabolic, and behavioral risk factors for type 2 diabetes at the end of the intervention (12mo) and after 1 year of follow-up (24mo).

ELIGIBILITY:
Inclusion Criteria:

* self-identify as American Indian
* BMI >=85th percentile for age and sex
* have at least one parent/primary caregiver (parent) willing to actively participate

Exclusion Criteria:

* diabetes
* any serious youth/parent health concerns that would interfere with participation
* plans to move out of the area during the study period

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 188 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change from 0 to 12 months in Body Mass Index (BMI) | 12 months
Change from 0 to 12 months in fasting insulin | 12 months

SECONDARY OUTCOMES:
Change from 0 to 12 months in BMI z-score | 12 months
Change from 0 to 12 months in waist circumference | 12 months
Change from 0 to 12 months in hemoglobin A1c | 12 months
Change from 0 to 12 months in fasting glucose | 12 months

OTHER OUTCOMES:
Change from 0 to 12 months in fruit/vegetable intake | 12 months
  Proportion consuming 5+ servings of fruits/vegetables daily
Change from 0 to 12 months in physical activity | 12 months
  Proportion engaging in 1+ hour of moderate-vigorous physical activity daily
Change from 0 to 12 months in screen time | 12 months
  Proportion watching 2 hours or less of screen time daily
Change from 0 to 12 months in sugary beverage intake | 12 months
  Proportion consuming 0 servings of sugary beverages daily
Participant engagement | 12 months
  Qualitative factors related to participant engagement
Program implementation | 12 months
  Qualitative factors related to program implementation
Potential for sustained delivery | 12 months
  Qualitative factors related to potential for sustained delivery

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Sauder, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Childrens Hospital Colorado, Aurora, Colorado, United States